CLINICAL TRIAL: NCT06884683
Title: A Phase II Study of Nivolumab Combined With Metformin in Pretreated Metastatic Renal Cell Carcinoma (mRCC) Patients. NivoMet TWINS-GU002 Study
Brief Title: Nivolumab Plus Metformin in Metastatic Renal Cell Carcinoma
Acronym: NivoMet
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, TORTORA GIAMPAOLO, Professor, Director of Medical Oncology and Comprehensive Cancer Center, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3209
Record Dates: First submitted 2023-03-14; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Metformin; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental (Experimental): nivolumab plus metformin Participants will receive nivolumab 240 mg e.v. every 14 days. Treatment will continue until progressive disease or discontinuation.
  Participants will receive metformin 500 mg orally twice a day. Treatment will continue until progressive disease or discontinuation.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Drug: metformin tablet 500 mg, 1 tablet twice a day (total dose 1000 mg daily), administered orally continuously
  +
  Biological: Nivolumab 240 mg via IV infusion every 14 days
  Other Names:
  Opdivo®
  Other Names: Nivolumab

SUMMARY:
Phase 2 single arm study that evaluated the addition of metformin to nivolumab in pre-treated metastatic renal cell carcinoma (mRCC) patients.

Primary aim: to investigate the efficacy of the combination of nivolumab+metformin in mRCC patients previously treated with VEGFR-TKI

Secondary aims:

* to assess the activity, safety and efficacy of the experimental combination
* to assess the quality of life of enrolled patients

Enrolled patients will received:

* nivolumab 240 mg e.v. every 14 day
* metformin 500 mg orally twice a day continuously Patients will be trated untill disease progression, or unexpected toxicity, whichever comes first

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Male and female aged 18 years and above
3. Histological confirmation of RCC with a clear cell component
4. Advanced or metastatic RCC
5. Measurable disease as defined by RECIST1.1criteria
6. Must have received at least one prior systemic treatment regimen in the advanced or metastatic setting, and must have evidence of progression on or after the last treatment regimen received
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2
8. Adequate bone marrow and chemistry values defined as:

   1. Hemoglobin ≥ 9.0 g/dL independent of transfusion
   2. Platelet count ≥100.000/μL
   3. Serum creatinine < 1.5 x ULN or a calculated creatinine clearance ≥ 40 mL/min
   4. Liver function:

   i. Serum bilirubin < 1.5 x ULN (except for patients with documented Gilbert's disease) ii. AST or ALT < 2.5 x ULN
9. Life expectancy of at least 6 months
10. WOCBP must use method(s) of contraception as determined to be acceptable by the principal investigator and sponsor during the study and for 23 weeks after last study drug administration.
11. Patients who are sexually active with WOCBP must be willing to use a method of birth control with adequate barrier protection as determined to be acceptable by the principal investigator and sponsor during the study and for 31 weeks after last study drug administration.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study:

1. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS). Any positive test for hepatitis B or hepatitis C virus indicating acute or chronic infection
2. Any active known or suspected autoimmune disease
3. Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days prior to the first dose of study drug. Inhaled steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease
4. Uncontrolled adrenal insufficiency
5. Evidence of active pneumonitis during screening, except for pulmonary fibrosis induced by prior thoracic irradiation
6. Dialitic patients
7. Diabetes mellitus
8. Any history of biguanide-based therapy within 1 year prior to enrollment
9. Current severe, uncontrolled systemic disease
10. Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class II-IV heart disease or cardiac ejection fraction measurement of < 50% at baseline
11. Other malignancy with a previous diagnosis within 5 years (with the exclusions of NMIBC, CIN).
12. Prior treatment with an anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
13. WOCBP who are pregnant or breastfeeding
14. Women with a positive pregnancy test at enrollment or prior to administration of study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
9-months PFS rate | 9 months after the last enrolled patient
  The percentage of patients without disease progression after 9 months from the start of therapy

SECONDARY OUTCOMES:
ORR | the ORR analysis will be performed after 12 months from the last patient enrolled
  objective response rate (percentage of patients with complete or partial response
median PFS | the PFS analysis will be performed after 12 months from the last patient enrolled
  median time of survival without disease progression
median OS | the OS analysis will be performed after 12 months from the last patient enrolled
  median time of overall survival
Adverse Events | AEs will be collected until 3 months from the discontinuation of the experimental therapy by the last patient enrolled
  description and rate of treatment-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Giampaolo Tortora, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (2):
- Italy (2):
  - Giampaolo Tortora, Roma
  - Francesca Primi, Viterbo

IPD SHARING:
Plan to Share IPD: No